CLINICAL TRIAL: NCT02155114
Title: Iron Homoeostasis in Inflammation: A Single Center Observational Cross-sectional Study
Brief Title: Iron Homoeostasis in Inflammation
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: EKNZ 2014-053; EKNZ 2014-053 (Other: Ethikkommission Nordwest- und Zentralschweiz)
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Inflammation; Bacterial Infections and Mycoses; Anemia, Iron-Deficiency; Iron Overload
Keywords: Hepcidins; Homeostasis; Iron/administration & dosage; Biological Markers/blood
MeSH Terms: conditions — Inflammation; Bacterial Infections and Mycoses; Anemia, Iron-Deficiency; Iron Overload

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood samples (serum and heparinized plasma)
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to survey iron storage levels and their prognostic consequences in the context of acute inflammation. The impact of iron substitution in inflammatory states is controversial. We hypothesize that iron substitution may influence outcome in patients in inflammatory states.

DETAILED DESCRIPTION:
* Background: Iron deficiency is frequently encountered in the elderly, after bleeding and in the context of neoplasia. Our 2013 pilot study showed that iron deficiency is a common problem in medical inpatients (13.7%) and that about 55% of these also showed signs of inflammation. The relevance of iron storage levels on clinical outcome in the presence of inflammation is conflicting. On the one hand, lack of iron prevents many viruses and bacteria, as well as other microorganisms, to reproduce and on the other hand the abundance of available iron stimulates hematopoiesis and reduces symptoms of iron deficiency.
* Methodology: We plan to enroll 1000-1500 patients with laboratory signs of inflammation during a period of six months and to analyze iron specific laboratory parameters twice during hospital stay. Additional laboratory analyses are planned for a smaller sample to portray the processes in iron homeostasis during inflammation.
* Significance: Contradicting evidence of forty and more years of scientific research backs current therapeutic practices in patients with inflammatory disease and iron deficiency. This study records prevalence of different iron storage states, mortality, morbidity and therapies in inflammatory states combined with iron deficiency and could very well be able to recommend a therapeutic regimen as well as limits for typically used laboratory parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18
* Hospitalized patient in internal medicine (≥ 24h)
* Evidence of an inflammatory state, determined as a C reactive protein (CRP) value >5 mg/l
* Written informed consent

Exclusion Criteria:

* History of terminal renal insufficiency in terms of dialysis or use of erythropoiesis-stimulating agents
* Pregnancy
* History of allogeneic stem cell transplantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive internal medicine inpatients with laboratory signs of inflammation
Sampling Method: Non-Probability Sample
Enrollment: 472 (Actual)
Dates: Start 2014-04; Primary Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of different iron states (normal iron states, iron deficiency and iron overload) in the context of acute inflammation | up to 8 days

SECONDARY OUTCOMES:
Correlation between iron states and clinical course of acute inflammation, mode of discharge and iron substitution | up to 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Balthasar L. Hug, MD, MBA, MPH, Principal Investigator — Division of Internal Medicine, University Hospital Basel, Switzerland
Locations (1):
- Basel University Hospital, Basel, Switzerland

REFERENCES:
- [Background] Hug BL, Tichelli A, Benkert P, Stirnimann G, Schifferli JA. Diagnosis and treatment of iron deficiency in medical inpatients at a Swiss tertiary university referral hospital: a retrospective observational cohort study of clinical practice. Swiss Med Wkly. 2013 Sep 6;143:w13847. doi: 10.4414/smw.2013.13847. eCollection 2013. PMID 24018778
- [Background] Thomas DW, Hinchliffe RF, Briggs C, Macdougall IC, Littlewood T, Cavill I; British Committee for Standards in Haematology. Guideline for the laboratory diagnosis of functional iron deficiency. Br J Haematol. 2013 Jun;161(5):639-648. doi: 10.1111/bjh.12311. Epub 2013 Apr 10. No abstract available. PMID 23573815
- [Background] Finberg KE. Unraveling mechanisms regulating systemic iron homeostasis. Hematology Am Soc Hematol Educ Program. 2011;2011:532-7. doi: 10.1182/asheducation-2011.1.532. PMID 22160085
- [Background] Drakesmith H, Prentice AM. Hepcidin and the iron-infection axis. Science. 2012 Nov 9;338(6108):768-72. doi: 10.1126/science.1224577. PMID 23139325
- [Background] Oppenheimer SJ. Iron and its relation to immunity and infectious disease. J Nutr. 2001 Feb;131(2S-2):616S-633S; discussion 633S-635S. doi: 10.1093/jn/131.2.616S. PMID 11160594